CLINICAL TRIAL: NCT00471393
Title: Double-blind Randomized Clinical Study on Topical Diclofenac Efficacy in Symptomatic Relief of Temporomandibular Degenerative Joint Disease in Women.
Brief Title: Topical Diclofenac Efficacy in Symptomatic Relief of Temporomandibular Degenerative Joint Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMW 5936; File #103090 Health Canada; Grant#2005-04; NCT00699647 (obsolete NCT alias)
Record Dates: First submitted 2007-05-07; First posted 2007-05-09 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Temporomandibular Degenerative Joint Disease
Keywords: TMJ; Osteoarthritis; Degenerative Joint disease
MeSH Terms: conditions — Osteoarthritis; Joint Diseases | interventions — Diclofenac; Dimethyl Sulfoxide; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 1.5% diclofenac in 45.5% DMSO (topical treatment)
Drug: 45.5% DMSO (topical placebo)

SUMMARY:
The use of a topical medication was compared to placebo to be applied over the symptomatic temporomandibular joint in women with the diagnosis of osteoarthritis of the temporomandibular joint(s).

The hypothesis is to investigate whether the use of a topical anti-inflammatory medication when compared to the placebo would decrease the pain of the affected joint and/or increased mouth opening.

DETAILED DESCRIPTION:
The purpose of this study is to measure the efficacy of topical diclofenac to topical placebo in the symptomatic relief of degenerative temporomandibular joint disease in a female population between the ages of 18-45 years of age.

Primary Objectives:

* To compare the efficacy of placebo and diclofenac topical PLO gel in terms of functional pain intensity of symptomatic temporomandibular degenerative joint disease in participants by comparing baseline measures obtained prior to commencement of the study, with the measurements obtained at 30, 60 and 90 days during the treatment intervention through the use of a Visual Analogue Scale (VAS).

Secondary Objectives:

* To compare the efficacy of placebo and diclofenac topical in PLO gel in terms of measurement of the range of motion of voluntary and assisted vertical jaw opening of symptomatic temporomandibular degenerative joint disease (TMDJD) in participants by comparing baseline measures obtained prior to commencement of the study, Time 0, through the use of a 100 mm ruler to measures obtained at 30, 60 and 90 days during the treatment intervention.
* To compare the efficacy of placebo and diclofenac in terms of effect on quality of life of symptomatic TMDJD in participants by comparing baseline measures obtained prior to commencement of the study, Time 0, to measures obtained after 90 consecutive days of treatment, utilizing a subsection of The Brief Pain Inventory Scale (BPI) which relates to quality of life.
* To compare the efficacy of placebo and diclofenac in terms of effect on pain intensity of symptomatic TMDJD in participants by comparing baseline measures obtained prior to commencement of the study, Time 0, to measures obtained after 90 consecutive days of treatment, utilizing a subsection of The Brief Pain Inventory Scale (BPI) (Cleeland & Ryan, 1994) which relates to pain intensity.
* To compare the efficacy of placebo and diclofenac topical PLO gel in terms of effect on disability on specific activities of daily living of TMDJD participants by comparing baseline measures obtained prior to the commencement of the study, Time 0, to that obtained after 90 consecutive day of treatment, utilizing The Pain Disability Index (PDI) (Bush & Harkin, 1995).

Tertiary Objectives

* To compare the adverse effects documented by the topical diclofenac group to those documented by the topical placebo group.
* To compare the amount of breakthrough medication used by the topical diclofenac group versus the placebo group in order to assess if the use of topical diclofenac reduces the amount of oral medication.
* To compare reasons for withdrawal from the study between topical placebo and topical diclofenac groups.

The null hypothesis is that there is no difference between the efficacy of topical diclofenac and topical placebo in the treatment of degenerative temporomandibular joint disease.

ELIGIBILITY:
Inclusion Criteria:

* A baseline score of ≥ 3.0 cm on a 10 cm measured VAS (Visual Analogue Scale) according to the criteria established by Collins et al. (Collins, Moore, & Mcquay, 1997) (for moderate and severe pain) required for participants prior to use of analgesics, in order to provide adequate sensitivity.
* Females from the ages of 18 to 45 years of age inclusive.
* Primary degenerative joint disease as diagnosed through radiographs utilizing volumetric cone beam computed tomographic images reformatted in axial, coronal, and sagittal views that will be assessed by an independent radiologist.

Exclusion Criteria:

* Nursing or expectant females or females planning on becoming pregnant.
* Participants not clearly diagnosed as having symptomatic degenerative joint disease.
* Participants having DJD secondarily to trauma, previous infection or general joint/muscle disease.
* Participants who have experienced adverse reactions to any of the components of the formulation used in the study.
* Participants who have evidence of periodontal disease, dental caries, oral pathology or infections of the oral cavity.
* Participants with a history of neuropathic pain in the orofacial region.
* Participants scheduled for surgery in the near future.
* Participants currently undergoing orthodontic treatment.
* Participants with a history of epilepsy, cardiovascular disease, renal disease/disorder, hepatic disease/disorder, glaucoma, bowel obstruction, urinary retention, diabetes, hypertension or orthostatic hypotension.
* Participants with a malignancy.
* Participants who are currently using topical preparations for palliative relief for their DJD.
* Participants with a baseline intensity of ≤ 3/10 on the VAS.
* Inability to understand English.
* Participants who have been wearing an occlusal splint ≤ 3 months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2006-05; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
1.To compare the efficacy of topical placebo and topical diclofenac in functional pain intensity at commencement of the study, Day 30, Day 60 and Day 90 through the use of VAS. | 90 days

SECONDARY OUTCOMES:
1.To compare the efficacy of topical placebo and topical diclofenac in voluntary and assisted vertical jaw opening through the use of a 100 mm ruler from commencement of the study, Day 30, Day 60 and Day 90. | 90 days
2.To compare the efficacy of topical placebo and topical diclofenac on the effect on quality of life by comparing measures at the commencement of the study to the end of treatment, through use of a subsection of The Brief Pain Inventory Scale (BPI). | 90 days
3.To compare the efficacy of topical placebo and topical diclofenac on pain intensity by comparing measures obtained at the commencement of the study, to those obtained at the end using a subsection of The Brief Pain Inventory Scale. | 90 days
4.To compare the efficacy of topical placebo and topical diclofenac on the disability on specific activities of daily living by comparing baseline measures, to that obtained at the end of treatment, utilizing The Pain Disability Index. | 90 days
5.To compare the adverse effects documented by the topical diclofenac group to those documented by the topical placebo group. | 90 days
6.To compare the amount of breakthrough medication used by the topical diclofenac group versus the topical placebo group in order to assess if the use of topical diclofenac reduces the amount of oral medication. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Norman Thie, BSc DDS MSc, Study Director — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Mason L, Moore RA, Edwards JE, Derry S, McQuay HJ. Topical NSAIDs for chronic musculoskeletal pain: systematic review and meta-analysis. BMC Musculoskelet Disord. 2004 Aug 19;5:28. doi: 10.1186/1471-2474-5-28. PMID 15317652
- [Background] Mason L, Moore RA, Edwards JE, Derry S, McQuay HJ. Topical NSAIDs for acute pain: a meta-analysis. BMC Fam Pract. 2004 May 17;5:10. doi: 10.1186/1471-2296-5-10. PMID 15147585
- [Background] Moore RA, Tramer MR, Carroll D, Wiffen PJ, McQuay HJ. Quantitative systematic review of topically applied non-steroidal anti-inflammatory drugs. BMJ. 1998 Jan 31;316(7128):333-8. doi: 10.1136/bmj.316.7128.333. PMID 9487165
- [Background] Roth SH, Shainhouse JZ. Efficacy and safety of a topical diclofenac solution (pennsaid) in the treatment of primary osteoarthritis of the knee: a randomized, double-blind, vehicle-controlled clinical trial. Arch Intern Med. 2004 Oct 11;164(18):2017-23. doi: 10.1001/archinte.164.18.2017. PMID 15477437
- [Background] Tugwell PS, Wells GA, Shainhouse JZ. Equivalence study of a topical diclofenac solution (pennsaid) compared with oral diclofenac in symptomatic treatment of osteoarthritis of the knee: a randomized controlled trial. J Rheumatol. 2004 Oct;31(10):2002-12. PMID 15468367
- [Background] Towheed TE. Pennsaid therapy for osteoarthritis of the knee: a systematic review and metaanalysis of randomized controlled trials. J Rheumatol. 2006 Mar;33(3):567-73. PMID 16511925